CLINICAL TRIAL: NCT06076759
Title: Intrathecal Dexmedetomidine Versus Intrathecal Morphine Inpatients Undergoing Cardiac Valve Replacement Surgeries: Effect on Postoperative Pain and Diaphragmatic Function
Brief Title: Intrathecal Dexmedetomidine Versus Intrathecal Morphine Inpatients Undergoing Cardiac Valve Replacement Surgeries
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Sara Usama Mohammed Rabie, Principle investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: Intrathecal analgesia
Record Dates: First submitted 2023-09-29; First posted 2023-10-11 (Actual); Last update posted 2023-10-11 (Actual); Status verified 2023-10

CONDITIONS: Cardiac Valve Disease
MeSH Terms: conditions — Heart Valve Diseases | interventions — Dexmedetomidine; Morphine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intrathecal morphine group (Group M): (Active Comparator): • Patients in this group will receive intrathecal morphine (0.5 mg diluted in I ml of normal saline) prior to induction of general anesthesia.
  Interventions: Drug: Intrathecal morphine or dexmedetomidine
- Intrathecal dexmedetomidine group (Group D): (Active Comparator): • Patients in this group will receive intrathecal dexmedetomidine (5 mcg diluted in 1 ml of normal saline) prior to induction of general anesthesia.
  Interventions: Drug: Intrathecal morphine or dexmedetomidine

INTERVENTIONS:
Drug: Intrathecal morphine or dexmedetomidine — Intrathecal injection
  Other Names: Morphine or dexmedetomidine

SUMMARY:
Comparison between the effects of intrathecal morphine versus intrathecal dexmedetomidine on analgesia and respiratory function, in open heart surgery.

DETAILED DESCRIPTION:
Postoperative pulmonary dysfunction is a well-recognized complication of open-heart surgeries. About 25% of patients who don't present with any severe impaired cardiac function reported to have significant pulmonary dysfunction for at least one week after operation. Many mechanisms could be accused of this dysfunction as respiratory mechanics failure by diaphragmatic paresis or paralysis, pain and muscle guarding, lung atelectasis, drains discomfort, etc.

although pain is the major concern of patients, but sometimes it may not get the proper attention, pain in open heart surgery origins mainly from the surgical incision which is here a median sternotomy the most commonly used approach and the easiest access to the heart region, however median sternotomy may significantly impedes the pulmonary function by the resultant pain of this procedure and cause morbidity and mortality by itself

ELIGIBILITY:
Inclusion Criteria:

- Cardiac patient scheduled for elective open heart valve replacement surgery.

Exclusion Criteria:

* • Patient refusal

  * Coagulation disorders
  * History of known allergy to the used drugs.
  * Combined procedures (e.gif combined with coronary artery bypass or aortic root surgeries).
  * If thoracotomy or min-sternotomy is planned for the surgery.
  * Re-do and emergency surgeries.
  * History of chronic chest diseases (COPD or IPF).
  * History of thoracotomy, pneumothorax, pneumomediastinum, phrenic nerve injury (as evident by the presence of paralysis of the ipsilateral hemidiaphragm when examined preoperatively).
  * Neuromuscular diseases.
  * Brain injuries.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-10-01 (Estimated); Primary Completion 2024-10-01 (Estimated); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
Total opioids consumption. | First 24 hour postoperatively
  Pain would be assessed subjectively by the patient using the numerical scale from 0 to 10 by the and boluses of fentanyl 1 mic/kg would be given when requested by the patient, then the total fentanyl consumption during the first 24h post operative would be calculated.

SECONDARY OUTCOMES:
Diaphragmatic function | First 24 hour postoperatively
  Chest ultrasonography for diaphragmatic function by measuring two parameters one is the diaphragmatic thickness and the other is diaphragmatic excursion at its largest echo, on both sides right and left, and by the same operator at three different settings, first is preoperative, second at time of spontaneous breathing trial postoperatively, and the last one is post extubation by 6 hours, and compare results to assess any diaphragmatic dysfunction even the subclinical one.

CONTACTS AND LOCATIONS:
Overall Officials: Hany Moustafa, Principal Investigator — Assiut University